CLINICAL TRIAL: NCT02246270
Title: Recurrent Urinary Tract Infections and Heparin: a Double-blind Randomized Trial (RUTIH Trial)
Brief Title: Recurrent Urinary Tract Infections and Heparin (RUTIH Trial)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8481
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravesical heparin (Experimental): Recurrent UTI subject receives intravesical heparin once every week for 6 weeks
  Interventions: Drug: Intravesical Heparin
- Placebo (Active Comparator): Recurrent UTI subject receives intravesical saline once every week for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intravesical Heparin — Heparin bladder instillation
  Other Names: Intravesical heparin bladder instillation
  Arms: Intravesical heparin
Other: Placebo — Intravesical saline
  Arms: Placebo

SUMMARY:
Urinary Tract Infections (UTIs) are the second most common infection in the body. UTIs account for five percent of all visits to primary care physicians. Many women who have had a UTI will develop recurring urinary tract infections. Recent studies suggest that some women who suffer from recurrent UTIs have urinary tracts that allow bacteria to adhere to it more readily than others. Women who suffered from bladder inflammation and recurrent UTIs were noted to have reduced UTIs and bladder inflammation with heparin bladder instillations. Heparin is a highly-sulfated glycosaminoglycan and stored within the secretory granules of mast cells and released only into the vasculature at sites of tissue injury. It has been proposed that, in addition to anticoagulation, the main purpose of heparin is defense at such sites against invading bacteria and other foreign materials. The central question the research is intended to answer is does Heparin bladder instillations decrease UTI rates in patients.

DETAILED DESCRIPTION:
Primary Objectives: The specific aims of this study are to 1) demonstrate that Heparin bladder instillations reduce the number of UTI episodes; 2) demonstrate Heparin bladder instillations increase median intervals between UTI; and 3) demonstrate that Heparin bladder instillations decrease urine inflammatory (NGAL) levels. Study Design: This study will be a randomized, double-blind, placebo-controlled trial of subjects treated for documented recurrent urinary tract infections with heparin bladder instillation versus sterile saline instillations. The study recruits women (n = 30) with 3 or more UTI episodes in one year from the patient population at The University of Oklahoma Health Sciences Center (OUHSC) and The University of Oklahoma-Tulsa (OU-Tulsa) and randomly assigns them to treatment as usual care with sterile saline instillation (n =15) or treatment as usual with heparin bladder instillations (n = 15). Subjects are given 6 weekly bladder instillations with interval follow-ups; the primary outcome measures are number of UTI episodes during the six month study period and a survival analysis assesses time to the next UTI. The usual care of this study is antibiotic treatment for UTI only. Urine samples will be collected at certain intervals. Analysis: We will seek a statistically significant difference of the recurrent UTI rate for 6 months between heparin instillation and sterile saline instillation group. Assuming Recurrent UTI rate of sterile saline bladder instillation is 2.3.3 UTI episodes per six months, a 35% reduction in the recurrent UTI rate is deemed significant based on previous literature. A sample size 30 (15 for each group) will achieve 60% power to detect a 35% reduction in recurrent UTI rate at a 0.05 significance level. Allowing for a 25% drop out, a total of 30 subjects will be required. Significance: Recurrent UTIs are challenging to manage, especially if microbiological results are equivocal. In women who suffer from frequent recurrences, daily antibiotic use is the most effective strategy for recurrent UTI prevention compared to daily cranberry pills, daily estrogen therapy, and acupuncture. However even with this traditional approach of continuous antibiotic for 6 to 12 months, the rate of UTI was only reduced during prophylaxis and the rate of UTI was unchanged after stopping antibiotic treatment. Increasing antibiotic resistance rates require immediate identification of innovative alternative prophylactic therapies. The lack of non-antibiotic therapies gives an opportunity to develop innovative strategies to decrease recurrent UTIs and decrease the burden of UTIs. This study will augment the current evidence available on the aggregate effects of a treatment that emphasizes the optimization of both antibiotic regimens and non-antibiotic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-85 with history of recurrent urinary tract infections.

  * Definition of Recurrent UTI: if experienced either more than 3 symptomatic UTI episodes in the past year (including the index infection) or 2 such episodes in the past 6 months.
  * Definition of UTI: >103 cfu/mL of a uropathogen in midstream urine culture from a woman experiencing more than 2 symptoms of cystitis (dysuria, urgency, frequency, suprapubic pain, or hematuria) or, in the absence of a culture, demonstration of pyuria on urinalysis and more than 2 urinary symptoms, as well as complete and rapid resolution of symptoms in response to antibiotic therapy for UTI.

Exclusion Criteria:

* Taking any anticoagulant such as warfarin sodium, heparin
* Taking any thrombolytic agent such as a tissue plasminogen activator or streptokinase
* Known aneurysm, thrombocytopenia, hemorrhagic disease, hemophilia, gastrointestinal ulceration, polyps, or diverticula
* Known hypersensitivity to heparin
* History of, or currently has neurogenic bladder, pelvic irradiation or chemical cystitis
* Presence of urethral, pelvic, or rectal carcinoma, Benign or malignant bladder tumors
* Tuberculous cystitis, urinary schistosomiasis
* Bladder or ureteral calculi, urethral or bladder obstruction, augmentation cystoplasty, cystectomy, supratrigonal denervation of the bladder (cystolysis), neurectomy, or implanted peripheral nerve stimulator that has affected bladder function; Microscopic hematuria as defined as > 5 red blood cells (RBC) /high power field at baseline visit without a negative workup within the last year
* Positive pregnancy test at the baseline visit, are pregnant or lactating, or are planning to become pregnant during the study period
* Have history of uterine, cervical or vaginal cancer during the past 3 years
* Clinically significant vaginitis at baseline visit

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in UTI rate at 6 months | 6 months
  Will measure change from baseline in UTI rate at 6 months using statistical methods

SECONDARY OUTCOMES:
Change from Baseline in median time to UTI recurrence at 6 months | 6 months
  Will measure change from baseline in median time to UTI recurrence at 6 months by statistical analysis

OTHER OUTCOMES:
Change from Baseline in NGAL levels at 6 months(NGAL) levels after Heparin treatment | 6 months
  Will measure change from baseline in NGAL levels at 6 months (NGAL) levels after Heparin treatment using statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jameca R. Price, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma-Tulsa OB/GYN Dept and OU-Physicians, Tulsa, Oklahoma, United States